CLINICAL TRIAL: NCT02902029
Title: A Phase II, Open-label, Randomized-controlled Trial Evaluating the Efficacy and Safety of a Sequencing Schedule of Cobimetinib Plus Vemurafenib Followed by Immunotherapy With an Anti- PD-L1 Antibody Atezolizumab for the Treatment in Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Brief Title: Evaluating the Efficacy and Safety of a Sequencing Schedule of Cobimetinib Plus Vemurafenib Followed by Immunotherapy With an Anti- PD-L1 Antibody in Patients With Unresectable or Metastatic BRAF V600 Mutant Melanoma
Acronym: ImmunoCobiVem
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Dirk Schadendorf, Prof. Dr. med., University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ImmunoCobiVem_2015
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Malignant Melanoma
Keywords: unresectable stage IIIB, IIIC, IV melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib; cobimetinib; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): After a 3 months run-in period with vemurafenib and cobimetinib [960 mg vemurafenib twice daily (BID), 28/0; 60 mg cobimetinib daily (QD), 21/7], all patients who do not show disease progression or definite treatment interruption (e.g. due to unacceptable toxicity) for more than 28 days will be randomized.
  Further treatment with vemurafenib and cobimetinib (960 mg vemurafenib BID, 28/0; 60 mg cobimetinib QD, 21/7).
  After progression of disease patients in Arm A will subsequently receive atezolizumab treatment (1200 mg/ q3w).
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib; Drug: Atezolizumab
- Arm B (Experimental): After a 3 months run-in period with vemurafenib and cobimetinib (960 mg vemurafenib BID, 28/0; 60 mg cobimetinib QD, 21/7), all patients who do not show disease progression or definite treatment interruption (e.g. due to unacceptable toxicity) for more than 28 days will be randomized.
  Further treatment with atezolizumab. Atezolizumab will be administered intravenously at a fixed dose of 1200 mg on day 1 of each 21 day-cycle.
  After progression of disease patients in Arm B will cross back to vemurafenib and cobimetinib treatment (960 mg vemurafenib BID, 28/0; 60 mg cobimetinib QD, 21/7).
  Interventions: Drug: Vemurafenib; Drug: Cobimetinib; Drug: Atezolizumab

INTERVENTIONS:
Drug: Vemurafenib — 960 mg vemurafenib BID until progression or unacceptable toxicity develops
Drug: Cobimetinib — 60 mg cobimetinib QD, 21/7 until progression or unacceptable toxicity develops
Drug: Atezolizumab — 1200 mg atezolizumab administered intravenously on day 1 of each 21 day-cycle. Will be given until progression or unacceptable toxicity develops

SUMMARY:
Most patients with locally advanced or metastatic tumors succumb to their disease. Thus, there is a substantial need for novel therapeutic strategies to improve the outcome for patients with advanced or metastatic melanoma. Targeting the the Ras/Raf signalling pathway by BRAF and MEK inhibition as well as targeting immunologic checkpoint control with an antiPD-L1 antibody have emerged as treatment option.

In this study the best timing for sequential use of both treatment options (BRAF/MEK inhibition and antiPD-L1 antibody) in patients with unresectable or metastatic BRAFV600 mutant melanoma will be assessed.

DETAILED DESCRIPTION:
At this time there is no experience concerning the sequencing strategy when using the two effective therapeutical approaches as targeting the Ras/Raf signalling pathway by BRAF and MEK inhibition or targeting immunologic checkpoint control with an antiPD-L1 antibody.

This is a prospective, open, multicenter, randomized phase II study in patients with unresectable or metastatic BRAFV600 mutant melanoma. In this study the scheduling of the treatment with a combined BRAF/MEK inhibition and the treatment with an anti-PD-L1 antibody will be assessed.

After a 3 months run-in period with vemurafenib and cobimetinib, all patients who did not show disease progression or treatment interruption for more than 28 days during run-in phase will be randomized in a 1:1 ratio:

* either to proceed vemurafenib and cobimetinib until disease progression and subsequently cross-over to atezolizumab treatment until disease progression (Arm A).
* or to receive the anti-PD-L1 antibody atezolizumab until disease progression and subsequently cross-back to vemurafenib and cobimetinib until disease progression (Arm B). In a translational research program tumor tissue, blood plasma and peripheral blood mononuclear cell will be analyzed to evaluate the biologic effects of treatment sequence on the molecular profile and biomarker expression in tissue and plasma.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial.
* Male or female patient being ≥18 years of age on day of signing informed consent.
* Histologically confirmed diagnosis of locally advanced, unresectable or metastatic melanoma AJCC (unresectable stage IIIB, IIIC, IVM1a, IVM1b, or IVM1c) without active or untreated brain metastases; all known CNS lesions must have been treated with stereotactic therapy or surgery at least 4 weeks prior to the first dose of trial treatment AND the patient must be without evidence of clinical or radiographic disease progression in the CNS for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms must have returned to baseline, the patient must have no evidence of new or enlarging brain metastases, and the patient must not have used steroids for at least 3 weeks prior to trial treatment.
* No previous therapy for the advanced or metastatic stage. Prior adjuvant therapy is permitted (e.g. Interferon, Interleukin-2-therapy, chemo- or radiotherapy). Prior adjuvant therapy has to be terminated (last dose) at least 28 days before enrolment. Patients who are in follow-up period of a clinical trial in adjuvant setting and progressing may be enrolled / randomized.
* Measurable disease, i.e., present with at least one measurable lesion per RECIST, version 1.1, for the definition of a measureable lesion.
* Presence of BRAF mutation (V600) in tumor tissue.
* Performance status of 0 or 1 on the ECOG Performance Scale.
* Adequate organ function.
* Adequate cardiac function.
* Able to take oral medications.
* Female subject of childbearing potential should have a negative pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Female patients of childbearing potential and male patients with partners of childbearing potential must agree to always use a highly effective form of contraception according to CTFG during the course of this study and for at least 6 months after completion of study therapy.

Exclusion Criteria:

* Use of any investigational or non-registered product within the 30 days before registration.
* Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to study Day 1.
* Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
* Prior therapy with a BRAF inhibitor (including but not limited to vemurafenib, dabrafenib, encorafenib and / or MEK inhibitor
* Prior major surgery.
* Known additional malignancy that is progressing or requires active treatment within 5 years prior to the study.
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* History of leptomeningeal metastases.
* History or current evidence of central serous retinopathy (CSR) or retinal vein occlusion (RVO) or predisposing factors to RVO or CSR.
* History of retinal degenerative disease.
* History of allogenic bone marrow transplantation or organ transplantation.
* History of Gilbert's syndrome.
* Impaired cardiovascular function or clinically significant cardiovascular diseases.
* Uncontrolled arterial hypertension despite medical treatment.
* Impairment of gastrointestinal function or gastrointestinal disease.
* Evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Active infection requiring systemic therapy.
* Positive test for Human Immunodeficiency Virus (HIV).
* Positive test for Hepatitis B or Hepatitis C.
* Known hypersensitivity reaction to any of the components of study treatment.
* Medical, psychiatric, cognitive or other conditions, including known alcohol or drug abuse.
* Patients having received a live, attenuated vaccine within 4 weeks prior to the first dose of trial treatment.
* Legal incapacity or limited legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2016-11; Primary Completion 2024-03 (Actual); Study Completion 2024-03 (Actual)

PRIMARY OUTCOMES:
Time to First Documented Disease Progression | 4 years
  Time to first documented disease progression (PFS1) defined as time from start of run-in phase (date of first intake of study drug) to first documented disease progression date according to RECIST v. 1.1. (PD1) or death by any cause, whichever occurs first.

SECONDARY OUTCOMES:
Time to Second Objective Disease Progression (PFS2) | 4 years
  Time to second objective disease progression (PFS2) defined as time from start of run-in phase (date of first intake of study drug) to second documented disease progression according to RECIST v. 1.1. (PD2) following randomization or death by any cause.
Adverse events according to CTCAE Version 4.03 criteria (Safety / Toxicity) | Until 90 days of discontinuation of dosing of the investigational product
  All adverse events according to CTCAE Version 4.03 criteria, and all serious adverse events regardless of causal relationship to the administration of the investigational agents will be assessed
Overall survival | 4 years
  Overall Survival (OS) of a patient defined as the time from start of run-in phase (date of first intake of study drug) until documented date of death
Overall survival 12 months | 1 year
  Overall survival rate at 12 months defined as the rate of patients alive 12 months after start of run-in phase (date of first intake of study drug)
Overall survival 24 months | 2 years
  Overall survival rate at 24 months defined as the rate of patients alive 24 months after start of run-in phase (date of first intake of study drug)
Overall survival 36 months | 3 years
  Overall survival rate at 36 months defined as the rate of patients alive 36 months after start of run-in phase (date of first intake of study drug)
Overall survival 48 months | 4 years
  Overall survival rate at 48 months defined as the rate of patients alive 48 months after start of run-in phase (date of first intake of study drug)
12-months disease control rate (DCR) | 1 year
  DCR is defined as the rate of patients showing complete response (CR) or partial response (PR) or stable disease (SD) at 12 months after start of run-in phase (date of first intake of study drug).
24-months disease control rate (DCR). | 2 years
  DCR is defined as the rate of patients showing complete response (CR) or partial response (PR) or stable disease (SD) at 24 months after start of run-in phase (date of first intake of study drug).
Rate of patients with progressive disease who could not cross-over to subsequent line of therapy due to deterioration of ECOG status or multiple and/or symptomatic brain metastases and/or leptomengial disease | 4 years
  * From vemurafenib + cobimetinib to atezolizumab (Arm A)
  * From atezolizumab to vemurafenib + cobimetinib (Arm B)
Time from first documented tumor progression until second documented tumor progression | 4 years
  PFS3 definded as time from first documented tumor progression (PD1) until second documented tumor progression (PD2) after randomization or death by any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (27):
- France (5):
  - Hôpital Ambroise-Paré, Boulogne-Billancourt
  - Hospital Claude Huriez, Lille
  - Hôpital de la Timone, Marseille
  - CHU de Nantes, Nantes
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
- Germany (20):
  - National Centre for Tumour Diseases (NCT), Heidelberg, Baden-Wurttemberg
  - SLK-Kliniken Heilbronn GmbH, Heilbronn, Baden-Wurttemberg
  - University Hospital Mannheim, Clinic for Dermatology, Mannheim, Baden-Wurttemberg
  - University Hospital Essen, Department of Dermatology, Skin Cancer Center, Essen, North Rhine-Westphalia
  - HELIOS Klinikum Erfurt, Erfurt, Thuringia
  - Charité-Universitätsmedizin Berlin, Berlin
  - Elbe Kliniken Stade - Buxtehude, Buxtehude
  - Universitätsklinikum Köln, Cologne
  - Universitätsklinik Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Universitäts-Hautklinik Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Gesellschaft für Klinische Forschung Ludwigshafen mbH, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Universitätsklinikum Mainz, Mainz
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum der Universität München, München
  - Universitätsklinikum Tübingen, Tübingen
  - Uniklinikum Würzburg, Würzburg
- "LAIKO" General Hospital of Athens, Athens, Greece
- Military Medical Academy, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No